CLINICAL TRIAL: NCT00863083
Title: Reducing Barriers to Behavior Change Among Youth With Pediatric Overweight and Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to poor enrollment.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Health System, Inc. (Other); Wisconsin Department of Health and Family Services (Other Government)
Responsible Party: Rachel Neff Greenley PhD/Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHW 08/101
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Pediatric Obesity; Pediatric Overweight
Keywords: pediatric obesity; pediatric overweight; multi-family group weight management intervention; financial rewards
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Multifamily group weight management intervention plus rewards for program attendance
  Interventions: Behavioral: Multifamily weight management intervention
- 2 (Active Comparator): Multifamily group weight management intervention plus rewards for attendance and goal attainment
  Interventions: Behavioral: Multifamily weight management intervention

INTERVENTIONS:
Behavioral: Multifamily weight management intervention — 8 week multifamily group weight management intervention incorporating behavioral health, nutrition, and activity disciplines.

SUMMARY:
The purpose of the study is to examine the extent to which two different reward systems implemented in the context of a multi-family pediatric weight management group differentially promote adoption of healthy eating and activity habits among overweight and obese 8-17 year old youth. Participants will be randomly assigned to one of two reward conditions: rewards for attendance only or rewards for attendance and goal attainment. We hypothesize that all participants will demonstrate significant increases in healthy nutritional choices and physical activity and significant reductions in sedentary activity from pre-intervention to post intervention. We expect that participants in attendance plus goal attainment reward condition will demonstrate significantly greater improvements than participants in the attendance only condition.

DETAILED DESCRIPTION:
Pediatric overweight and obesity are significant public health concerns, and group based interventions incorporating behavioral, nutrition, and activity disciplines have showed modest success in improving youth health and weight status. The role of financial rewards in encouraging attendance at weight management sessions and acquisition of healthy eating and activity habits is not well understood in the context of pediatric weight management, however. Behavior theory suggests that positive reinforcement can increase the frequency of desirable behaviors. As such, the primary goal of the study is to evaluate the role of different reinforcement systems in increasing healthy nutritional choices, increasing physical activity, and decreasing sedentary activity among youth participating in a multifamily group based pediatric overweight/obesity intervention program. An additional aim of the study is to evaluate the role of different levels of rewards in decreasing BMI among youth participating in a multifamily group based pediatric overweight/obesity intervention program. Participants will be randomly assigned to one of two different reward conditions: Condition A (rewards for attendance only) and Condition A+G (rewards for attendance and goal attainment).

Up to 80 participants will be recruited to participate. Eligibility criteria include patient age 8-17 years, patient with public insurance managed by Children's Community Health Network, English speaking patient and parent, and patient body mass index at or above the 85th percentile for age and sex. Exclusion criteria include: significant patient developmental or cognitive delay, or concurrent involvement in another formal weight management program.

Pre and post intervention assessments of anthropometric, psychosocial, nutritional, and physical fitness variables will be conducted, and participants will complete 8 weekly multi-family group-based weight management intervention sessions involving psychology, physical therapy, and dietitian disciplines. Following this intensive phase, families will follow up on a quarterly basis for one year. Families will receive financial rewards for attending program sessions (Conditions A and A+G) and for completing behavioral monitoring assignments (Condition A+G).

ELIGIBILITY:
Inclusion Criteria:

* patient age 8-17 years
* patient with public insurance managed by Children's Community Health Network
* English speaking patient and parent
* patient body mass index at or above the 85th percentile for age and sex
* parent or legal guardian willing to participate

Exclusion Criteria:

* significant patient developmental or cognitive delay
* concurrent involvement in another formal weight management program.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
dietary habits | pre, post, quarterly follow ups
physical and sedentary activity | pre, post, quarterly follow ups

SECONDARY OUTCOMES:
body mass index | pre, post, quarterly follow ups
participant satisfaction | post intevention

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Neff Greenley, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Children's Hosptial of Wisconsin, Milwaukee, Wisconsin, United States